CLINICAL TRIAL: NCT00000341
Title: Pharmacokinetics and Bioavailability of Liquid vs Tablet Buprenorphine
Brief Title: Evaluation of Liquid vs. Tablet Buprenorphine - 6
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-3-0010-6; Y01-3-0010-6
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-08

CONDITIONS: Opioid-Related Disorders
Keywords: opioid dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to evaluate the steady-state pharmacokinetics and bioavailability of buprenorphine sublingual tablets vs. sublingual solution.

ELIGIBILITY:
Inclusion Criteria:

M/F ages 21-50. Meet DSM-IV criteria for opioid dependence. Agree to conditions of the study and sign informed consent.

Exclusion Criteria:

Psychiatric disorder that requires medication therapy. History of seizures. Pregnant and/or nuring women. Dependence on ETOH or benzodiazepines or other sedative/hypnotics. Acute hepatitis. Other medical condtions that deem participation to be unsafe.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1
Dates: Start 1996-08; Study Completion 2000-08 (Actual)

PRIMARY OUTCOMES:
Subjective and observer rater physiological effects of bup

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States